CLINICAL TRIAL: NCT00353561
Title: Diabetes Mellitus and Vulvovaginal Candidiasis: Prevalence of Infection and Its Rationale Management
Brief Title: Diabetes Mellitus and Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Responsible Party: Ravinder Goswami, All India Institute of Medical Sciences, New Delhi 110029
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHN/Adhoc/23/2003-2004
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus; Vulvovaginal Candidiasis
MeSH Terms: conditions — Diabetes Mellitus; Candidiasis, Vulvovaginal | interventions — boric acid; Fluconazole

ARMS (2):
- 1, Boric acid (Active Comparator): 600 mg vaginal pessaries for 14 days
  Interventions: Drug: Boric
- 2, Fluconazole (Other)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Boric — Gelatin capsules filled with 600 mg of boric acid
  Arms: 1, Boric acid
Drug: Fluconazole — 150 mg oral fluconazole gives once in 14 days
  Arms: 2, Fluconazole

SUMMARY:
Clinical and mycological response to oral fluconazole and boric acid suppositories was assessed in patients with diabetes mellitus and vulvovaginal candidiasis.

DETAILED DESCRIPTION:
A high proportion of vulvovaginal candidiasis is due to C.glabrata that responds poorly to fluconazole therapy. We assessed the clinical relief and mycological cure in response to oral fluconazole and boric acid suppositories in patients with diabetes mellitus and vulvovaginal candidiasis given in a Randomized trial. Fluconazole was given in standard oral single dose (150 mg) fluconazole and boric acid vaginal suppositories was given in dose of 600 mg/daily for 14 uninterrupted days.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with diabetes mellitus attending Endocrine OPD of All India Institute of Medical Sciences and in whom the diagnosis of vulvovaginal candidiasis was based on presence of clinical signs and symptoms and growth of Candida species on culture of high vaginal swab (HVS).

Exclusion Criteria:

* Patients with vaginal discharge in whom Candida growth was not detected on fungal culture were excluded.
* Subjects also excluded were those with pregnancy,
* Sexually inactive girls,
* Age > 65 years, renal failure and steroid therapy.
* Patients who did not give consent for pelvic examination,
* Those who were treated for any kind of vaginal discharge during the past three months and who did not comply with boric acid therapy or did not report on 15th day for repeat examination excluded.

Ages: 18 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Mycological cure on the 15th day of therapy and defined as the absence of Candida growth on fungal culture of high vaginal swab | 15 days

SECONDARY OUTCOMES:
Relief in clinical symptoms and signs of vulvovaginal candidiasis including vaginal discharge, pruritus, burning sensation and vaginal congestion | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Goswami, DM, Principal Investigator — All India Institute of Medical Sciences New Delhi, 110029, India
Locations (1):
- Dr Ravinder Goswami, Delhi, National Capital Territory of Delhi, India

REFERENCES:
- See also: PMID: 17692922 and 17259500, J Infection 2007 and Diabetes Care 2007 — http://www.ncbi.nlm.nih.gov/sites/entrez